CLINICAL TRIAL: NCT02146469
Title: Study on Effectiveness of 2-dose Live Attenuated Varicella Vaccine
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Shanghai Municipal Center for Disease Control and Prevention (Other)
Collaborators: Shanghai Institute Of Biological Products (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SH2012VAR
Record Dates: First submitted 2014-05-21; First posted 2014-05-23 (Estimated); Last update posted 2014-05-23 (Estimated); Status verified 2014-05

CONDITIONS: Varicella
Keywords: varicella vaccination
MeSH Terms: conditions — Chickenpox | interventions — Chickenpox Vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- None varicella vaccine history (Experimental): 2 doses with an 3 months interval
  Interventions: Biological: 2 doses with an 3 months interval
- 1 year after first dose (Experimental): A second dose with an 1 year interval
  Interventions: Biological: A second dose with an 1 year interval
- 3 years after first dose (Experimental): A second dose with an 3 year interval
  Interventions: Biological: A second dose with an 3 year interval
- 5 years after first dose (Experimental): A second dose with an 5 year interval
  Interventions: Biological: A second dose with an 5 year interval
- Testing group for conbined immunization (Experimental): 1 dose Varicella vaccine and 1 dose MMR given at the same time
  Interventions: Biological: 1 dose Varicella vaccine and 1 dose MMR given at the same time
- Control group for conbined immunization (Placebo Comparator): 1 dose MMR
  Interventions: Biological: 1 dose MMR

INTERVENTIONS:
Biological: 2 doses with an 3 months interval — varicella vaccination
  Arms: None varicella vaccine history
Biological: A second dose with an 1 year interval — varicella vaccine
  Arms: 1 year after first dose
Biological: A second dose with an 3 year interval — varicella vaccine
  Arms: 3 years after first dose
Biological: A second dose with an 5 year interval — varicella vaccine
  Arms: 5 years after first dose
Biological: 1 dose Varicella vaccine and 1 dose MMR given at the same time — varicella vaccine and MMR
  Arms: Testing group for conbined immunization
Biological: 1 dose MMR — MMR
  Arms: Control group for conbined immunization

SUMMARY:
The objective of the study is as follows:

1. To know the antibody level during different interval after received 1 dose varicella vaccine.
2. To know safety and effectiveness of received 2 doses varicella vaccine with different interval.
3. To know safety and effectiveness of received varicella vaccine and MMR at the same time.

To achieve that, this study selects children with specific varicella vaccine history, gives 1 or 2 doses varicella vaccine, collects blood specimens and makes a follow-up visit after vaccination.

All blood specimens will be tested by a third-party detection institution.

ELIGIBILITY:
Inclusion Criteria:

* Aged 1 to 7
* Without a previous history of varicella
* With an axillary temperature ≤37.5℃ at the time of vaccination
* Appropriate varicella vaccination history
* With guardian signing the informed consent and available for clinical observation

Exclusion Criteria:

* Hypersensitive to any active substance of the vaccine including excipients and antibiotics
* With acute illness, severe or acute attack of chronic illness or fever
* With immunodeficiency or weakened immune system or being treated with immunosuppressant drugs
* Suffering a brain disease, uncontrolled epilepsy or progressive nerve system disease
* With a family or personal history of seizure, chronic illness, epilepsy or allergy
* With unknown immunization history or unable to follow the immunization schedule of EPI
* Received any vaccine within 4 weeks or willing to receive any vaccine in 1 month
* With hemorrhagic tendency or prolonged period of bleeding
* Received whole blood, plasma or immunoglobulin within 5 months
* Received systemic antibiotics or antiviral treatment for acute illness within 7 days
* With an axillary temperature ≥38℃ within 3 days
* Participating in another clinical trial
* Any situation that might influence the consequence of the clinical trial

Ages: 1 Year to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1200 (Estimated)
Dates: Start 2012-12; Primary Completion 2014-06 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Seroconversion rate and GMCs after varicella vaccination | 35-42 days after each dose vaccination

SECONDARY OUTCOMES:
The incidence of Adverse Events Following Immunization | 30 days after each dose vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Xiaodong Sun, Study Director — Shanghai Municipal Center for Disease Control and Prevention
Locations (1):
- Shanghai municipal center for disease control and prevention, Shanghai, Shanghai Municipality, China